CLINICAL TRIAL: NCT01917955
Title: Cardiac MRI in Ischemic Stroke Study
Acronym: CaMriSS
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Center for Stroke Research Berlin (Other); Cardiology and Angiology, Elisabeth Hospital, Essen, Germany (Unknown)
Responsible Party: Principal Investigator, Karl Georg Haeusler, MD, Charite University, Berlin, Germany
Other Study IDs: CaMriSS_CSB; EA4/073/10 (Other: Charité Ethics Committee)
Record Dates: First submitted 2012-08-07; First posted 2013-08-07 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-11

CONDITIONS: Stroke
Keywords: MRI
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this prospective single-center trial is to compare the safety and diagnostic value of contrast medium-enhanced cardiac magnetic resonance imaging and transesophageal echocardiography in patients with acute ischemic stroke.

DETAILED DESCRIPTION:
Primary safety objective: Contrast medium-enhanced cardiac magnetic resonance imaging is safe in patients with acute ischemic stroke. Primary outcome: The diagnostic value of contrast medium-enhanced cardiac magnetic resonance imaging is comparable to transesophageal echocardiography in patients with acute ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute ischemic stroke detected by brain magnetic resonance imaging.

Exclusion Criteria:

* Known atrial fibrillation or cardiac source of embolism
* Severe aphasia
* Acute infection or chronic inflammation
* Severe arteriosclerosis or stenosis of brain-supplying arteries
* Contraindications for magnetic resonance imaging or transesophageal echocardiography.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Overall, 103 patients with acute ischemic stroke detected by brain magnetic resonance imaging will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2012-01; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of contrast medium-enhanced cardiac magnetic resonance imaging to detect echocardiography-proven cardiac sources of embolism in patients with acute ischemic stroke. | < 1 week after ischemic stroke

SECONDARY OUTCOMES:
Rate of unrecognised myocardial infarction detected by late gadolinium-enhanced cardiac MRI in patients with acute ischemic stroke. | < 1 week after ischemic stroke

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Matthias Endres, MD, Study Chair — Center for Stroke Research Berlin; Karl Georg Haeusler, MD, Principal Investigator — Center for Stroke Research Berlin
Locations (2):
- Germany (2):
  - Charité, Universitätsmedizin Berlin, Campus Benjamin Franklin, Berlin
  - Elisabeth Hospital, Essen

REFERENCES:
- [Derived] Haeusler KG, Wollboldt C, Bentheim LZ, Herm J, Jager S, Kunze C, Eberle HC, Deluigi CC, Bruder O, Malsch C, Heuschmann PU, Endres M, Audebert HJ, Morguet AJ, Jensen C, Fiebach JB. Feasibility and Diagnostic Value of Cardiovascular Magnetic Resonance Imaging After Acute Ischemic Stroke of Undetermined Origin. Stroke. 2017 May;48(5):1241-1247. doi: 10.1161/STROKEAHA.116.016227. Epub 2017 Apr 14. PMID 28411261